CLINICAL TRIAL: NCT02139410
Title: Insulin Like Growth Factor 1 and Risks of Sarcopenia and Mortality in Patients With Cognitive Impairment
Brief Title: IGF-1, Sarcopenia and Mortality: a Cohort Study in Patient With Cognitive Impairment
Acronym: ISAAC
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Vincenzo Gianturco, MD, University of Roma La Sapienza
Other Study IDs: IGF-001
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-09

CONDITIONS: Cognitive Impairment; Insulin-like Growth Factor 1
Keywords: sarcopenia; mortality
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IGF-1 1st and 2nd quartile: Reduction of IGF-1 serum value in a cohort of patients with cognitive impairment
  Interventions: Procedure: IGF-1 serum value
- IGF-1 3rd and 4rd quartile: Reduction of IGF-1 serum value in a cohort of patients with cognitive impairment
  Interventions: Procedure: IGF-1 serum value

INTERVENTIONS:
Procedure: IGF-1 serum value — Evaluation of IGF-1 serum value at baseline, 24 and 48 months

SUMMARY:
Insulin-like growth factor 1 (IGF)-1 is an important neuromyotrophic hormone. Disregulation of this hormone has been reported to influence the genesis of cognitive impairment and dementia in the elderly patients. We analyzed the possible link between IGF-1 and risk of Sarcopenia and Mortality in a cohort of elder patients with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cognitive impairment (MMSE < 24)
* Age > 65 ys

Exclusion Criteria:

* Diagnosis of pancreatic disorders
* Diagnosis of acromegaly
* Diagnosis of GH-related disorders
* Recent bone fractures or immobility before the enrollment (3 months)
* Cancer

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive patients were enrolled from orthopedics clinic (IRCCS Galeazzi Milan) and geriatric day service (Sapienza University of Rome)
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2008-06; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
IGF-1 reduction in patients with sarcopenia | baseline, 24 months, 48 months
  IGF-1 reduction could be linked to sarcopenia in patients with cognitive impairment

SECONDARY OUTCOMES:
IGF-1 reduction and mortality in patients with cognitive impairment | baseline, 24 months, 48 months
  IGF-1 could be an independent risk factor for mortality in patients with cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Gianturco, MD, Principal Investigator — University of Roma La Sapienza
Locations (2):
- Italy (2):
  - IRCCS Galeazzi, Milan, Italy
  - Sapienza University of Rome, Rome, Italy